CLINICAL TRIAL: NCT01170156
Title: Fluid Leakage Past Tracheal Tube Cuff : Effect of Suctioning Manoeuvre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Roanne (Other)
Responsible Party: Véronique BOURRACHAUT, CH de Roanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010REACHR01; 2010-A00539-30 (Other: AFSSAPS)
Record Dates: First submitted 2010-07-22; First posted 2010-07-27 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Deep Sedation; Respiration, Artificial
Keywords: deep sedation; respiratory resuscitation; Hi-Lo Evac tube; suctioning manoeuvre
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Hi-Lo Evac tube (Mallinckrodt Inc, USA) (Instilled blue dye) — The cuff pressure will be first checked and reset at 30 cm H2O if needed. Next, blue dye will be instilled just above the cuff through the lumen ending in the subglottic area of the Hi-Lo Evac tube. Then a suctioning manoeuvre will be performed with a suction pressure of - 400 mbar through a 16 French suction catheter. Thereafter, a fiberoptic bronchoscopy will be performed, looking for the presence of blue dye in the trachea and/or the bronchi.
  Other Names: Hi-Lo Evac tube (Mallinckrodt Inc, USA); Blue dye 2.5% (Guerbet, France)

SUMMARY:
The leakage of oropharyngeal secretions around high-volume low-pressure tracheal tube cuffs is usually considered as a major risk factor for bacterial tracheal colonization and subsequent development of ventilator-associated pneumonia. The rate of leakage around the cuff is related to the pressure differential across the cuff, namely the difference between the pressure of the subglottic fluid above the cuff and the tracheal pressure under the cuff. Consequently, positive end-expiratory pressure (PEEP) improves the sealing around the cuff towards fluid leakage. However, this preventive effect of PEEP is compromised during prolonged mechanical ventilation by tracheal suctioning manoeuvre, which may enhance fluid leakage, by decreasing tracheal pressure. Indeed, in a benchtop model, a suctioning manoeuvre, without disconnection of the ventilator, induced a constant fluid leakage past a high-volume low-pressure tracheal tube cuff when performed with a high level of suction pressure (- 400 mbar) and a large size of suction catheter size (16 French).

DETAILED DESCRIPTION:
This clinical study aims to confirm these experimental data in patients under mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* intubated with a Hi-Lo Evac tube since less than 48 hours
* under continuous sedation
* written consent signed

Exclusion Criteria:

* hemodynamic instability
* allergy of blue dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Presence of blue dye in the trachea and/or the bronchi after the suctioning manoeuvre. | 48 hours after the beginning of the mechanical ventilation
  The cuff pressure will be first checked and reset at 30 cm H2O if needed. Next, blue dye will be instilled just above the cuff through the lumen ending in the subglottic area of the Hi-Lo Evac tube. Then a suctioning manoeuvre will be performed with a suction pressure of - 400 mbar through a 16 French suction catheter. Thereafter, a fiberoptic bronchoscopy will be performed, looking for the presence of blue dye in the trachea and/or the bronchi.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BEURET, MD, Principal Investigator — CH de Roanne
Locations (1):
- CH de Roanne, Roanne, France

REFERENCES:
- [Derived] Beuret P, Philippon B, Fabre X, Kaaki M. Effect of tracheal suctioning on aspiration past the tracheal tube cuff in mechanically ventilated patients. Ann Intensive Care. 2012 Nov 7;2(1):45. doi: 10.1186/2110-5820-2-45. PMID 23134813